CLINICAL TRIAL: NCT03396445
Title: A Phase 1 Study of MK-5890 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Brief Title: Study of Boserolimab (MK-5890) as Monotherapy and in Combination With Pembrolizumab (MK-3475) in Adults With Advanced Solid Tumors (MK-5890-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5890-001; MK-5890-001 (Other: MSD); 2017-004550-41 (EudraCT Number)
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Pharmacokinetics; Solid Tumor; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1); Programmed Cell Death Receptor Ligand 2 (PD-L2); PD-1; PDL1; PD-L1; PD-L2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Pemetrexed; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Arm 1 Boserolimab 2 mg Q3W (Experimental): Participants receive boserolimab 2 mg via intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1 Boserolimab 7 mg Q3W (Experimental): Participants receive boserolimab 7 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1 Boserolimab 20 mg Q3W (Experimental): Participants receive boserolimab 20 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1 Boserolimab 70 mg Q3W (Experimental): Participants receive boserolimab 70 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1 Boserolimab 200 mg Q3W (Experimental): Participants receive boserolimab 200 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1 Boserolimab 700 mg Q3W (Experimental): Participants receive boserolimab 700 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 1a Boserolimab 30 mg Q3W (Endometrial) (Experimental): Participants with endometrial cancer receive boserolimab 30 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab
- Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W (Experimental): Participants receive separate IV infusions of boserolimab 2 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W (Experimental): Participants receive separate IV infusions of boserolimab 7 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W (Experimental): Participants receive separate IV infusions of boserolimab 20 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W (Experimental): Participants receive separate IV infusions of boserolimab 70 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W (Experimental): Participants receive separate IV infusions of boserolimab 200 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) (Experimental): Participants with triple-negative breast cancer (TNBC) receive separate IV infusions of boserolimab 30 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) (Experimental): Participants with endometrial cancer receive separate IV infusions of boserolimab 30 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) (Experimental): Participants with endometrial cancer receive separate IV infusions of boserolimab 30 mg and pembrolizumab 400 mg. Boserolimab was administered once every 6 weeks (Q6W) on Day 1 of each cycle for a total of up to approximately 4 cycles (up to approximately 6 months). Pembrolizumab is administered once Q6W on Day 1 of each cycle for a total of up to approximately 18 cycles (up to approximately 27 months). Each cycle is 6 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab
- Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) (Experimental): Participants with non-small cell lung cancer (NSCLC) receive separate IV infusions of boserolimab 30 mg, pembrolizumab 200 mg, pemetrexed 500 mg/m^2, and carboplatin area under the curve (AUC) 5 mg/mL/min. Boserolimab is administered once Q3W on Day 1 of each cycle for a total of up to approximately 8 cycles (up to approximately 6 months). Pembrolizumab and pemetrexed are administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Carboplatin is administered once Q3W on Day 1 of each cycle for a total of up to approximately 4 cycles (up to approximately 3 months). Each cycle is 3 weeks long.
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) (Experimental): Participants with TNBC receive separate IV infusions of boserolimab 30 mg, pembrolizumab 400 mg, and nab-paclitaxel 100 mg/m^2. Boserolimab and pembrolizumab are administered once Q6W on Day 1 of each cycle for a total of up to approximately 18 cycles (up to approximately 27 months). Nab-paclitaxel is administered on a 3-weeks on/1-week off schedule every 28 days (Days 1, 8, 15, 29, and 36 of odd-numbered cycles and Days 1, 15, 22, and 29 of even-numbered cycles). Each cycle is 6 weeks long
  Interventions: Drug: Boserolimab; Biological: Pembrolizumab; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Boserolimab — IV infusion
  Other Names: MK-5890
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W; Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W; Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W; Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W; Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W; Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC); Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial); Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial); Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC); Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Drug: Pemetrexed — IV infusion
  Other Names: ALIMTA®
  Arms: Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC)
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
  Arms: Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC)
Drug: Nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
  Arms: Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of boserolimab (MK-5890) when administered alone and in combination with pembrolizumab (MK-3475) in adults. Boserolimab monotherapy or boserolimab plus pembrolizumab combination therapy will be administered in adults with advanced solid tumors, including endometrial cancer, for up to 35 administrations (approximately 2 years). The safety and pharmacokinetics of boserolimab when administered with pembrolizumab, pemetrexed and carboplatin in adults with non-squamous non-small cell lung cancer (NSCLC) and boserolimab when administered with pembrolizumab and nab-paclitaxel in adults with triple-negative breast cancer (TNBC) will also be assessed.

DETAILED DESCRIPTION:
Participants receiving boserolimab monotherapy who experience disease progression may be eligible to switch to receiving boserolimab plus pembrolizumab combination therapy at an eligible dose for up to 35 cycles (approximately 2 years) at the discretion of the Investigator and approval of the Sponsor.

Per protocol, pharmacokinetic (PK) outcome measures will not be analyzed separately for the switch-over treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Arms 1 & 2: Histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and has received or been intolerant to all treatment known to confer clinical benefit
* Arm 3: Histologically or cytologically confirmed diagnosis of stage IV (M1a or M1b per current American Joint Committee on Cancer criteria) non-squamous NSCLC
* Arm 4: Triple-negative breast cancer (TNBC) that is locally recurrent, inoperable, not previously treated with chemotherapy, and which cannot be treated with curative intent OR metastatic disease not previously treated with chemotherapy
* Measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by the local site investigator/radiologist. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Male participants must agree to use adequate contraception during the treatment period and for at least 120 days after the last dose of boserolimab or pembrolizumab OR 180 days after the last dose of chemotherapeutic agents and refrain from donating sperm during this period
* Female participants must not be pregnant or breastfeeding and agree to follow use adequate contraception during the treatment period and for at least 120 days after the last dose of boserolimab or pembrolizumab OR 180 days after the last dose of chemotherapeutic agents
* Submit an evaluable baseline tumor sample for analysis (either a newly obtained or archival tumor sample)

Exclusion Criteria:

* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Clinically active central nervous system metastases and/or carcinomatous meningitis
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody (mAb) and/or other components of the study treatment
* Active infection requiring systemic treatment
* History of interstitial lung disease
* History of (noninfectious) pneumonitis that required steroids or current pneumonitis
* Symptomatic ascites or pleural effusion
* Previously had a stem cell or bone marrow transplant
* Previously had a solid organ transplant
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) except vitiligo or resolved childhood asthma/atopy
* Known human immunodeficiency virus (HIV) and/or active and acute Hepatitis B or C infections
* Not fully recovered from any effects of major surgery without significant detectable infection
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) before the first dose of study treatment, or has not recovered to Grade ≤1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier
* Expected to require any other form of antineoplastic therapy while participating in this study
* On chronic systemic steroid therapy in excess of replacement doses (e.g., exceeding 10 mg/day of prednisone equivalent), or on any other form of immunosuppressive medication
* Regular user (including "recreational use") of any illicit drugs at the time of signing informed consent, or has a recent history (within the last year) of substance abuse (including alcohol), as determined by the treating investigator. Participants who use cannabis for medicinal purposes or to treat specific symptoms will not be excluded unless it is being abused in the opinion of the treating investigator
* Received a live-virus vaccine within 28 days before the first dose of study treatment
* Currently participating and receiving study treatment in a study of an investigational agent or has participated and received study treatment in a study of an investigational agent or has used an investigational device within 28 days before the first dose of study treatment

Additional Exclusion Criteria for Participants in Arm 3:

* Has received radiation therapy to the lung that is >30 Gray (Gy) within 6 months before the first dose of study treatment
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Is unable or unwilling to take folic acid or vitamin B12 supplementation

Additional Exclusion Criteria for Participants in Arm 4:

* Has a known history of hypersensitivity or allergy to nab-paclitaxel or any of its components
* Has neuropathy ≥Grade 2
* Has a history of class II-IV congestive heart failure or myocardial infarction within 6 months of randomization
* Has received previous treatment with immune checkpoint inhibitor(s) (eg, Programmed Cell Death Receptor 1 (PD-1)/PD-L1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (18):
- United States (3):
  - University of South Alabama, Mitchell Cancer Institute ( Site 0020), Mobile, Alabama
  - Florida Cancer Specialists ( Site 0002), Sarasota, Florida
  - The West Clinic, P.C. ( Site 0021), Germantown, Tennessee
- Chile (2):
  - FALP-UIDO ( Site 0502), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0501), Santiago, Region M. de Santiago
- Israel (3):
  - Soroka Medical Center-Oncology ( Site 0012), Beersheba
  - Hadassah Ein Kerem Medical Center ( Site 0010), Jerusalem
  - The Chaim Sheba Medical Center - Oncology Institute ( Site 0001), Ramat Gan
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 0003), Amsterdam, North Holland
  - Erasmus MC ( Site 0031), Rotterdam, South Holland
- South Korea (2):
  - Seoul National University Hospital-Internal Medicine ( Site 0702), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 0701), Seoul
- Spain (4):
  - Hospital Universitario Quiron Madrid ( Site 0043), Pozuelo de Alarcón, Madrid
  - Instituto Catalan de Oncologia - ICO ( Site 0044), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 0041), Madrid
  - Centro Integral Oncologico Clara Campal START Madrid ( Site 0040), Madrid
- Taiwan (2):
  - National Taiwan University Hospital-Oncology ( Site 0801), Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0802), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, pharmacokinetic (PK) outcome measures were not analyzed separately for the switch-over treatment arms.
Groups:
- Arm 1 Boserolimab 2 mg Q3W: Participants received boserolimab 2 mg via intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long
- Arm 1 Boserolimab 7 mg Q3W: Participants received boserolimab 7 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1 Boserolimab 20 mg Q3W: Participants received boserolimab 20 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1 Boserolimab 70 mg Q3W: Participants received boserolimab 70 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1 Boserolimab 200 mg Q3W: Participants received boserolimab 200 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1 Boserolimab 700 mg Q3W: Participants received boserolimab 700 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1a Boserolimab 30 mg Q3W (Endometrial): Participants with endometrial cancer received boserolimab 30 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W: Participants received separate IV infusions of boserolimab 2 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W: Participants received separate IV infusions of boserolimab 7 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W: Participants received separate IV infusions of boserolimab 20 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W: Participants received separate IV infusions of boserolimab 70 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W: Participants received separate IV infusions of boserolimab 200 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC): Participants with triple-negative breast cancer (TNBC) received separate IV infusions of boserolimab 30 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial): Participants with endometrial cancer received separate IV infusions of boserolimab 30 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial): Participants with endometrial cancer received separate IV infusions of boserolimab 30 mg and pembrolizumab 400 mg. Boserolimab was administered once Q6W on Day 1 of each cycle for a total of up to approximately 4 cycles (up to approximately 6 months). Pembrolizumab was administered once every 6 weeks (Q6W) on Day 1 of each cycle for a total of up to approximately 18 cycles (up to approximately 27 months). Each cycle was 6 weeks long.
- Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC): Participants with non-small cell lung cancer (NSCLC) received separate IV infusions of boserolimab 30 mg, pembrolizumab 200 mg, pemetrexed 500 mg/m^2, and carboplatin area under the curve (AUC) 5 mg/mL/min. Boserolimab was administered once Q3W on Day 1 of each cycle for a total of up to approximately 8 cycles (up to approximately 6 months). Pembrolizumab and pemetrexed were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Carboplatin was administered once Q3W on Day 1 of each cycle for a total of up to approximately 4 cycles (up to approximately 3 months). Each cycle was 3 weeks long.
- Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC): Participants with TNBC received separate IV infusions of boserolimab 30 mg, pembrolizumab 400 mg, and nab-paclitaxel 100 mg/m^2. Boserolimab and pembrolizumab were administered once Q6W on Day 1 of each cycle for a total of up to approximately 18 cycles (up to approximately 27 months). Nab-paclitaxel was administered on a 3-weeks on/1-week off schedule every 28 days (Days 1, 8, 15, 29, and 36 of odd-numbered cycles and Days 1, 15, 22, and 29 of even-numbered cycles). Each cycle was 6 weeks long.
- Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 2 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 2 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 7 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 2 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 20 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 7 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 20 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 20 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 70 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 20 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 200 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 20 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 200 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 70 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W: Qualified participants who received boserolimab 200 mg via IV infusion in Arm 1 but experienced disease progression switched over to receive separate IV infusions of boserolimab 200 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
- Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W: Qualified participants who received boserolimab 30 mg via IV infusion in Arm 1a but experienced disease progression switched over to receive separate IV infusions of boserolimab 30 mg and pembrolizumab 200 mg. Boserolimab and pembrolizumab were administered once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years) after switch-over. Each cycle was 3 weeks long.
Period: Treatment Period
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Started | 3 | 3 | 6 | 3 | 9 | 2 | 14 | 3 | 3 | 4 | 7 | 14 | 31 | 15 | 14 | 10 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 3 | 3 | 6 | 3 | 8 | 2 | 14 | 3 | 3 | 3 | 7 | 14 | 30 | 15 | 13 | 10 | 41 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 3 | 9 | 2 | 14 | 3 | 3 | 4 | 7 | 12 | 30 | 14 | 13 | 8 | 19 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 1 | 1 | 3 | 2 | 5 | 3 | 3 | 3 | 7 | 12 | 28 | 14 | 10 | 8 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized by Mistake without Study Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease, Switched Over to Boserolimab + Pembrolizumab Combination Treatment | 1 | 1 | 5 | 2 | 5 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Switch-over Period
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Started (Per protocol, participants who experience disease progression in boserolimab monotherapy Arms 1 or 1a had the option, at the investigator's discretion and after consultation with the Sponsor, to switch over to boserolimab + pembrolizumab combination therapy at an eligible dose.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 9
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 1 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol, baseline characteristics were not analyzed separately for the switch-over period.
Groups:
- Arm 1 Boserolimab 2 mg Q3W: Participants received boserolimab 2 mg via IV infusion once Q3W on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long.
- Arm 1 Boserolimab 7 mg Q3W: Participants received boserolimab 7 mg via intravenous (IV) infusion once every 3 weeks (Q3W) on Day 1 of each cycle for a total of up to approximately 35 cycles (up to approximately 2 years). Each cycle was 3 weeks long
- Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial): Participants with endometrial cancer received separate IV infusions of boserolimab 30 mg and pembrolizumab 400 mg. Boserolimab was administered once Q6W on Day 1 of each cycle for a total of up to approximately 4 cycles (up to approximately 6 months). Pembrolizumab was administered once Q6W on Day 1 of each cycle for a total of up to approximately 18 cycles (up to approximately 27 months). Each cycle was 6 weeks long.
- Total: Total of all reporting groups
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 9 | 2 | 14 | 3 | 3 | 4 | 7 | 14 | 31 | 15 | 14 | 10 | 41 | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (18.9) | 57.3 (18.0) | 57.0 (15.8) | 54.0 (15.7) | 61.6 (14.2) | 61.0 (2.8) | 71.6 (5.7) | 44.7 (15.6) | 50.0 (24.3) | 61.5 (6.2) | 59.9 (7.2) | 55.1 (16.1) | 50.4 (13.3) | 64.6 (7.1) | 68.5 (9.5) | 61.9 (9.4) | 51.7 (11.8) | 57.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 5 | 2 | 14 | 2 | 0 | 1 | 7 | 10 | 31 | 15 | 14 | 6 | 41 | 155
  Male | 1 | 2 | 4 | 1 | 4 | 0 | 0 | 1 | 3 | 3 | 0 | 4 | 0 | 0 | 0 | 4 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 11 | 14
  Not Hispanic or Latino | 3 | 3 | 6 | 3 | 5 | 2 | 14 | 3 | 3 | 4 | 6 | 14 | 26 | 14 | 13 | 9 | 30 | 158
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 15 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
  White | 3 | 3 | 6 | 3 | 6 | 2 | 13 | 3 | 3 | 4 | 7 | 13 | 30 | 13 | 14 | 10 | 26 | 159
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last) of Boserolimab
Description: AUC0-last was defined as the area under the concentration versus time curve for boserolimab from 0 to the time of the last quantifiable concentration in serum. Samples were taken predose and at specified times postdose to determine the AUC0-last of boserolimab.
  PK collection time frames include: Arms 1, 2 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 5, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 1a, 2a, 2b, 3 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 2c and 4 (Cycle = 6 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15, 22 of Cycle 1, and predose on Day 1 of Cycle 2.
Time Frame: Predose Day 1 Cycle 1 and at designated timepoints up to Day 1 Cycle 2
Population: All participants who complied with the protocol sufficiently to ensure that the data was likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available AUC0-last data from ≥1 study treatment. As pre-specified in the protocol, PK outcomes were not analyzed separately for the Switch-over Arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 3 | 1 | 3 | 3 | 8 | 2 | 14 | 2 | 3 | 2 | 7 | 14 | 30 | 15 | 11 | 10 | 40
day*μg/mL | 0.761 (179) | 7.61 (NA) — Method of dispersion could not be estimated due to n=1. | 44.4 (28.6) | 150 (14.2) | 469 (42.9) | 918 (21.4) | 44.4 (51.7) | 0.816 (20.8) | 3.9 (117) | 26.1 (38.5) | 84.5 (192) | 646 (16.3) | 41.5 (109) | 44.9 (68.6) | 47.5 (58.5) | 41.6 (44.5) | 62.9 (57.8)

2. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. A DLT was defined as any of the following events: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia requiring a platelet transfusion; Nonhematologic adverse event (AE) Grade ≥3, with exceptions; Grade 3 or 4 nonhematologic laboratory abnormality; Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity; Treatment-related toxicity resulting in study drug discontinuation during the DLT evaluation period; Missing >25% of any study drug during the DLT evaluation period due to a treatment-related AE; or Grade 5 toxicity. The number of participants who experienced one or more DLTs is reported.
Time Frame: Up to 21 days in Cycle 1
Population: All participants in Arms 1, 1a, 2, 2a, 2b, 2c, and Switch-over Arms who received ≥1 dose of study treatment and who were observed for DLTs for up to 21 days following the first dose of study treatment in Cycle 1. As pre-specified in the protocol, DLTs were analyzed separately for the Switch-over Arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 8 | 2 | 14 | 3 | 3 | 3 | 7 | 14 | 30 | 15 | 13 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 9
Participants | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Number of Participants With One or More AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced one or more AEs is reported.
Time Frame: Up to approximately 78 months
Population: All participants in Arms 1, 1a, 2, 2a, 2b, 2c, and Switch-over Arms who received ≥1 dose of study treatment. As pre-specified in the protocol, safety data were analyzed separately for the Switch-over Arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 8 | 2 | 14 | 3 | 3 | 3 | 7 | 14 | 30 | 15 | 13 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 9
Participants | 3 | 3 | 6 | 3 | 8 | 2 | 14 | 3 | 3 | 3 | 7 | 14 | 30 | 15 | 13 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 8

4. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to 23 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 8 | 2 | 14 | 3 | 3 | 3 | 7 | 14 | 30 | 15 | 13 | 1 | 1 | 2 | 3 | 2 | 2 | 2 | 1 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2

5. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 3 Weeks (AUC0-3w) of Boserolimab
Description: AUC0-3w was defined as the area under the concentration versus time curve for boserolimab from 0 to 3 weeks in serum. Samples were taken predose and at specified times postdose to determine the AUC0-3w of boserolimab.
  PK collection time frames include: Arms 1, 2 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 5, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 1a, 2a, 2b, 3 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 2c and 4 (Cycle = 6 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15, 22 of Cycle 1.
Time Frame: Predose Day 1 Cycle 1 and at designated timepoints up to Day 1 Cycle 2
Population: All participants who complied with the protocol sufficiently to ensure that the data was likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available AUC0-3w data from ≥1 study treatment. As pre-specified in the protocol, PK outcomes were not analyzed separately for the Switch-over Arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 3 | 1 | 3 | 3 | 8 | 2 | 14 | 2 | 3 | 2 | 7 | 14 | 30 | 15 | 11 | 10 | 40
day*μg/mL | 1.79 (111) | 7.77 (NA) — Method of dispersion could not be estimated due to n = 1 | 44.4 (28.6) | 155 (7.85) | 531 (28.1) | 1060 (0.434) | 44.3 (54) | 1.2 (22) | 6.69 (47.5) | 28.1 (50.8) | 142 (63.3) | 661 (16.4) | 49.9 (41.3) | 50.5 (34.2) | 48.1 (42.5) | 42.2 (41.5) | 60.4 (39.5)

6. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to 6 Weeks (AUC0-6w) of Boserolimab
Description: AUC0-6w was defined as the area under the concentration versus time curve for boserolimab from 0 to 6 weeks in serum. Samples were taken predose and at specified times postdose to determine the AUC0-6w of boserolimab. As pre-specified in the protocol, different arms had different sampling schedules and cycle lengths and therefore AUC0-6w was not analyzed for all Arms; AUC0-6w was only analyzed for Arms 2c and 4 which had 6-week cycles.
Time Frame: Arms 2c and 4 (Cycle = 6 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15, 22 of Cycle 1, and predose on Day 1 Cycle 2
Population: All participants in Arms 2c and 4 who complied with the protocol sufficiently to ensure that the data was likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available AUC0-6w data from ≥1 study treatment. As pre-specified in the protocol, PK outcomes were not analyzed separately for the Switch-over Arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 11 | 40
day*μg/mL | 55 (49.2) | 68.3 (45.4)

7. Secondary Outcome: Minimum Concentration (Cmin) of Boserolimab
Description: Cmin of boserolimab was defined as the minimum concentration of boserolimab observed in serum. Samples were taken predose and at specified times postdose to determine the Cmin of boserolimab.
  PK collection time frames include: Arms 1, 2 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 5, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 1a, 2a, 2b, 3 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 2c and 4 (Cycle = 6 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15, 22 of Cycle 1, and predose on Day 1 of Cycle 2.
Time Frame: Predose Day 1 Cycle 1 and at designated timepoints up to Day 1 Cycle 2
Population: All participants who complied with the protocol sufficiently to ensure that the data was likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available Cmin data from ≥1 study treatment. As pre-specified in the protocol, PK outcomes were not analyzed separately for the Switch-over Arms.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 3 | 2 | 3 | 2 | 5 | 1 | 13 | 2 | 2 | 3 | 5 | 13 | 26 | 15 | 10 | 9 | 36
μg/mL | NA (NA) — For all 3 participants, plasma concentrations of boserolimab were below the limits of quantitation. | 0.0689 (0.0975) | 0.421 (0.103) | 3.55 (0.573) | 15.5 (8.08) | 24.3 (NA) — Method of dispersion could not be estimated due to n = 1 | 0.617 (0.498) | NA (NA) — For all 2 participants, plasma concentrations of boserolimab were below the limits of quantitation. | 0.0283 (0.0400) | 0.0629 (0.0575) | 3.55 (3.37) | 16.2 (5.14) | 0.721 (0.505) | 0.610 (0.499) | 0.126 (0.258) | 0.471 (0.473) | 0.158 (0.340)

8. Secondary Outcome: Maximum Concentration (Cmax) of Boserolimab
Description: Cmax of boserolimab was defined as the maximum concentration of boserolimab observed in serum. Samples were taken predose and at specified times postdose to determine the Cmax of boserolimab.
  PK collection time frames include: Arms 1, 2 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 5, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 1a, 2a, 2b, 3 (Cycle = 3 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15 of Cycle 1, and predose on Day 1 of Cycle 2; Arms 2c and 4 (Cycle = 6 weeks): Predose, at start & end of infusion on Day 1 Cycle 1, Days 2, 3, 8, 15, 22 of Cycle 1, and predose on Day 1 of Cycle 2.
Time Frame: Predose Day 1 Cycle 1 and at designated timepoints up to Day 1 Cycle 2
Population: All participants who complied with the protocol sufficiently to ensure that the data was likely to exhibit the effects of treatment, according to the underlying scientific model, and who had available Cmax data from ≥1 study treatment. As pre-specified in the protocol, PK outcomes were not analyzed separately for the Switch-over Arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 3 | 1 | 3 | 3 | 8 | 2 | 14 | 2 | 3 | 2 | 7 | 14 | 30 | 15 | 11 | 10 | 40
μg/mL | 1.15 (175) | 3.32 (NA) — Method of dispersion could not be estimated due to n = 1 | 8.16 (28.6) | 21.6 (22) | 67.8 (23.1) | 105 (8.71) | 7.24 (46.7) | 0.656 (5.08) | 1.75 (5.75) | 4.9 (39) | 26.9 (37) | 83.2 (16.6) | 7.89 (70.2) | 8.68 (24.6) | 8.27 (37.4) | 7.44 (37.3) | 9.39 (33.2)

9. Secondary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. As pre-specified in the protocol, ORR was analyzed for participants treated with boserolimab when used as monotherapy in Arm 1a, in combination with pembrolizumab in Switch-over Arm 1a and Arms 2a, 2b, and 2c, or in combination with pembrolizumab + nab-paclitaxel in Arm 4. Per protocol, ORR was not analyzed in Arms 1, 2, or 3. The percentage of participants who experienced a CR or PR, as assessed by the investigator, is reported.
Time Frame: Up to approximately 78 months
Population: All participants in Arm 1a, 2a, 2b, 2c, 4, and Switch-over Arm 1a with a baseline scan who demonstrated measurable disease by investigator assessment, and who were administered at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
Number analyzed (Participants) | 14 | 30 | 15 | 13 | 41 | 9
Percentage of Participants | 7.1 [0.2 to 33.9] | 20.0 [7.7 to 38.6] | 13.3 [1.7 to 40.5] | 0.0 [0.0 to 24.7] | 53.7 [37.4 to 69.3] | 11.1 [0.3 to 48.2]
Statistical Analysis 1: Comparison: Arm 1a Boserolimab 30 mg Q3W (Endometrial) vs Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial); Difference in percentage of participants who experienced a CR or PR (Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W [Endometrial] - Arm 1a Boserolimab 30 mg Q3W [Endometrial]); Test type: Other; Difference in Percent = 6.2, 95% CI 2-sided [-21.2 to 32.8] — Comparison based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Arm 1a Boserolimab 30 mg Q3W (Endometrial) vs Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial); Difference in percentage of participants who experienced a CR or PR (Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W [Endometrial] - Arm 1a Boserolimab 30 mg [Endometrial]); Test type: Other; Difference in Percentage = -7.1, 95% CI 2-sided [-32.1 to 17.2] — Comparison based on Miettinen & Nurminen method
Statistical Analysis 3: Comparison: Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) vs Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial); Difference in percentage of participants who experienced a CR or PR (Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W [Endometrial] - Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W [Endometrial]); Test type: Other; Difference in Percentage = 13.3, 95% CI 2-sided [-11.7 to 38.4] — Comparison based on Miettinen & Nurminen method

10. Secondary Outcome: Arm 3: Number of Participants Who Experienced a DLT
Description: DLTs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. A DLT was defined as any of the following events: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia requiring a platelet transfusion; Nonhematologic adverse event (AE) Grade ≥3, with exceptions; Grade 3 or 4 nonhematologic laboratory abnormality; Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity; Treatment-related toxicity resulting in study drug discontinuation during the DLT evaluation period; Missing >25% of any study drug during the DLT evaluation period due to a treatment-related AE; or Grade 5 toxicity. The number of participants who experienced one or more DLTs in Arm 3 is reported
Time Frame: Up to 21 days in Cycle 1
Population: All participants in Arm 3 who received ≥1 dose of study treatment and who were observed for DLTs for up to 21 days following the first dose of study treatment in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC)
Number analyzed (Participants) | 10
Participants | 0

11. Secondary Outcome: Arm 4: Number of Participants Who Experienced a DLT
Description: DLTs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. A DLT was defined as any of the following events: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia requiring a platelet transfusion; Nonhematologic adverse event (AE) Grade ≥3, with exceptions; Grade 3 or 4 nonhematologic laboratory abnormality; Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity; Treatment-related toxicity resulting in study drug discontinuation during the DLT evaluation period; Missing >25% of any study drug during the DLT evaluation period due to a treatment-related AE; or Grade 5 toxicity. The number of participants who experienced one or more DLTs in Arm 4 is reported.
Time Frame: Up to 28 days in Cycle 1
Population: All participants in Arm 4 who received ≥1 dose of study treatment and who were observed for DLTs for up to 28 days following the first dose of study treatment in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 41
Participants | 1

12. Secondary Outcome: Arm 3 and 4: Number of Participants With One or More AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Arms 3 and 4 who experienced one or more AEs is reported.
Time Frame: Up to 57 months
Population: All participants in Arms 3 or 4 who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 10 | 41
Participants | 10 | 41

13. Secondary Outcome: Arm 3 and 4: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Arms 3 or 4 who discontinued study treatment due to an AE is reported.
Time Frame: Up to 27 months
Population: All participants in Arms 3 or 4 who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC)
Number analyzed (Participants) | 10 | 41
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Up to approximately 78 months
Description: Serious & other AEs: all participants who received ≥1 dose of study drug. All-Cause Mortality (ACM): all enrolled participants. Per protocol, progression of cancer under study was not considered an AE unless related to study drug; MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. ACM and AEs are reported according to the treatment received by the participant at the time of the event.
Arm/Group | Arm 1 Boserolimab 2 mg Q3W | Arm 1 Boserolimab 7 mg Q3W | Arm 1 Boserolimab 20 mg Q3W | Arm 1 Boserolimab 70 mg Q3W | Arm 1 Boserolimab 200 mg Q3W | Arm 1 Boserolimab 700 mg Q3W | Arm 1a Boserolimab 30 mg Q3W (Endometrial) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 1/6 | 1/3 | 3/9 | 2/2 | 5/14 | 3/3 | 3/3 | 4/4 | 7/7 | 12/14 | 29/31 | 14/15 | 10/14 | 8/10 | 18/41 | 0/1 | 1/1 | 2/2 | 2/3 | 1/2 | 2/2 | 0/2 | 1/1 | 6/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/6 | 0/3 | 1/8 | 1/2 | 2/14 | 1/3 | 0/3 | 1/3 | 1/7 | 3/14 | 11/30 | 2/15 | 0/13 | 9/10 | 13/41 | 0/1 | 0/1 | 1/2 | 1/3 | 0/2 | 2/2 | 0/2 | 0/1 | 3/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 8/8 | 2/2 | 14/14 | 3/3 | 3/3 | 3/3 | 7/7 | 14/14 | 30/30 | 15/15 | 13/13 | 10/10 | 40/41 | 1/1 | 1/1 | 2/2 | 3/3 | 2/2 | 2/2 | 2/2 | 1/1 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Boserolimab 2 mg Q3W (N=3) | Arm 1 Boserolimab 7 mg Q3W (N=3) | Arm 1 Boserolimab 20 mg Q3W (N=6) | Arm 1 Boserolimab 70 mg Q3W (N=3) | Arm 1 Boserolimab 200 mg Q3W (N=8) | Arm 1 Boserolimab 700 mg Q3W (N=2) | Arm 1a Boserolimab 30 mg Q3W (Endometrial) (N=14) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W (N=7) | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W (N=14) | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) (N=30) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) (N=15) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) (N=13) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) (N=10) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) (N=41) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=3) | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W (N=9)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Boserolimab 2 mg Q3W (N=3) | Arm 1 Boserolimab 7 mg Q3W (N=3) | Arm 1 Boserolimab 20 mg Q3W (N=6) | Arm 1 Boserolimab 70 mg Q3W (N=3) | Arm 1 Boserolimab 200 mg Q3W (N=8) | Arm 1 Boserolimab 700 mg Q3W (N=2) | Arm 1a Boserolimab 30 mg Q3W (Endometrial) (N=14) | Arm 2 Boserolimab 2 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 7 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 20 mg Q3W + Pembrolizumab 200 mg Q3W (N=3) | Arm 2 Boserolimab 70 mg Q3W + Pembrolizumab 200 mg Q3W (N=7) | Arm 2 Boserolimab 200 mg Q3W + Pembrolizumab 200 mg Q3W (N=14) | Arm 2a Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (TNBC) (N=30) | Arm 2b Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W (Endometrial) (N=15) | Arm 2c Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W (Endometrial) (N=13) | Arm 3 Boserolimab 30 mg Q3W + Pembrolizumab 200 mg Q3W + Pemetrexed + Carboplatin (NSCLC) (N=10) | Arm 4 Boserolimab 30 mg Q6W + Pembrolizumab 400 mg Q6W + Nab-paclitaxel (TNBC) (N=41) | Switch-over Arm 1 Boserolimab 2 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1 Boserolimab 7 mg Q3W To Boserolimab 2 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 7 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 20 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=3) | Switch-over Arm 1 Boserolimab 70 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 20 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 70 mg + Pembrolizumab 200 mg Q3W (N=2) | Switch-over Arm 1 Boserolimab 200 mg Q3W To Boserolimab 200 mg + Pembrolizumab 200 mg Q3W (N=1) | Switch-over Arm 1a Boserolimab 30mg Q3W (Endometrial) To Boserolimab 30mg + Pembrolizumab 200mg Q3W (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 18 (54) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (60) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 10 (65) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 2 (2) | 5 (10) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 5 (6) | 2 (2) | 0 (0) | 3 (3) | 13 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 6 (10) | 1 (1) | 5 (9) | 18 (45) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 12 (16) | 4 (5) | 5 (7) | 5 (8) | 22 (33) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 9 (13) | 2 (2) | 2 (2) | 1 (1) | 11 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 1 (2) | 5 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 12 (13) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 6 (7) | 9 (10) | 18 (20) | 4 (6) | 3 (3) | 6 (7) | 25 (41) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 1 (1) | 2 (2) | 6 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 3 (3) | 17 (25) | 0 (0) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 2 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 4 (5) | 10 (11) | 4 (5) | 5 (6) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 6 (6) | 0 (0) | 2 (2) | 2 (4) | 14 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 11 (23) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 5 (5) | 0 (0) | 3 (3) | 2 (7) | 15 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 5 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 15 (38) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 13 (35) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 3 (5) | 10 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 3 (10) | 9 (16) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 2 (3) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 17 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 3 (4) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 1 (3) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (4) | 12 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 16 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIth nerve paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 3 (3) | 13 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 3 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 20 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 7 (7) | 11 (11) | 2 (2) | 2 (2) | 2 (2) | 22 (29) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 17 (27) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 5 (5) | 4 (5) | 1 (1) | 3 (3) | 8 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial prior to submission. Any information identified by the Sponsor as confidential must be deleted prior to submission. This confidentiality does not include efficacy and safety results. The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT03396445/Prot_SAP_000.pdf